CLINICAL TRIAL: NCT04767022
Title: A Prospective, Multicenter, Randomized Controlled Trials to Evaluate the Safety and Effectiveness of Genoss® DCB Versus SeQuent® Please NEO in Patients with Coronary In-stent Restenosis (ISR)
Brief Title: Compare the Safety and Effectiveness of Genoss® DCB and SeQuent® Please NEO in Chinese Patients with Coronary ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-DS1001-C
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: In-Stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genoss® DCB (Experimental): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: Paclitaxel Coated PTCA Balloon Catheter(Genoss® DCB)
- SeQuent® Please NEO (Active Comparator): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: Paclitaxel Coated PTCA Balloon Catheter(SeQuent® Please NEO)

INTERVENTIONS:
Device: Paclitaxel Coated PTCA Balloon Catheter(Genoss® DCB) — Drug Coated Balloon
  Arms: Genoss® DCB
Device: Paclitaxel Coated PTCA Balloon Catheter(SeQuent® Please NEO) — Drug Coated Balloon
  Arms: SeQuent® Please NEO

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Genoss® DCB by demonstrating non-inferiority in patients with in-stent restenosis (ISR) compared with a product of the same category (Sequent® Please NEO).

The experimental group was treated with Genoss® DCB, and the control group was treated with SeQuent® Please NEO.

In this study, the end point of 9 months after procedure was used as the main endpoint to evaluate the effectiveness of Paclitaxel coated PTCA balloon catheter. The safety of the catheter was evaluated by cardiovascular adverse events.

DETAILED DESCRIPTION:
In a randomized controlled trials to compare with the same-category medical device (Sequent® Please NEO), 224 patients with in-stent restenosis (ISR) were recruited from a total of 13 institutions, and the enrolled subjects were 1: 1 through randomization. The ratio was assigned to the test group(Genoss® DCB) and the control group(SeQuent® Please NEO), and each of the test or control devices was assigned to receive the procedure.

All patients were followed up 30 days, 6 months, 9 months, 1 year and 2 years after procedure, and angiographic follow-up was performed 9 months after procedure.

ELIGIBILITY:
Inclusion Criteria:

Subject related inclusion criteria

* Age≥18 years old & ≤80 years old.
* Patients with stable angina pectoris, unstable angina pectoris, stable acute myocardial infarction or confirmed silent myocardial ischemia.
* Patients who can understand the purpose of the study and voluntarily participate in and sign informed consent.
* It is suitable for patients undergoing percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).

Desease related inclusion criteria

* The target lesions were in stent restenosis: Mehran type I, II and III stenosis.
* The stenosis rate of target lesion diameter was more than 70%, or more than 50%, accompanied by objective evidence of ischemia (such as stress electrocardiogram, myocardial perfusion imaging, FFR, etc.)
* The reference vessel diameter of the target lesion was 2.0-4.0 mm, and the target lesion length was less than or equal to 26 mm.
* It is expected that no more than two drug balloons will be used in each subject, and each target lesion can be covered by one drug balloon.
* At most 2 primary lesions need interventional treatment, and the distance from the target lesion is more than or equal to 10 mm, and can be successfully treated before the intervention of the target lesion.

Exclusion Criteria:

Subject related exclusion criteria

* A woman who is pregnant, lactating, or planning a pregnancy.
* Patients with cardiogenic shock, acute infection, known bleeding or coagulation disorder, or history of cerebral hemorrhage, subarachnoid hemorrhage, active peptic ulcer and gastrointestinal bleeding within 3 months before operation.
* Patients who are known to be allergic to aspirin, clopidogrel, ticagrelor, heparin, contrast agent, paclitaxel, or have contraindications to aspirin, clopidogrel or ticagrelor.
* Patients with acute myocardial infarction within 1 week before operation.
* Patients with Takayasu arteritis.
* Left ventricular ejection fraction ≤ 30%.
* Acute or chronic renal insufficiency (serum creatinine > 2.0mg/dl or 178 μ mol / L).
* Patients with life expectancy less than 1 year.
* Patients participating in clinical trials of other drugs or medical devices.
* According to the researcher's judgment, the patient's clinical condition is not suitable for this study, or the patient is expected to be unable to complete the follow-up study according to the protocol.

Disease related exclusion criteria

* The target lesion was total occlusion (Mehran type IV).
* The target and non target lesions were left main artery lesions.
* The target lesions were ostial, pontine and bifurcated lesions with branch diameter ≥ 2.5mm.
* Three vessel disease requiring treatment.
* More than 3 lesions (including target lesions and non target lesions) need to be treated in target vessels.
* ISR lesions intervened within 6 months before operation.
* Angiography confirmed thrombus in the target vessel.
* The target vessel is severely calcified, tortuous and angulated, so it is expected that the drug balloon catheter will not pass successfully.
* The lesions that could not be pre dilated successfully were grade C or above dissection after pre dilation, or residual stenosis > 30%, or TIMI blood flow < grade III.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss after procedure | at 9 months after procedure
  In-segment late lumen loss between test group(Genoss DCB) and control group(Sequent Please) evaluated by quantitiative coronary analysis in patients with ISR

SECONDARY OUTCOMES:
Device-oriented compoiste endpoint (DOCE) | at 30 days, 6 months, 9 months, 12 months and 24 months after procedure
  DOCE is defined as a composite of cadiac death, target vessel-related myocardial infarction (TV-MI), and ischemia-driven target lesion revascularization (ID-TLR)
Patient-oriented composite endpoint (POCE) | at 30 days, 6 months, 9 months, 12 months, and 24 months after procedure
  POCE is defined as a composite of all-cause death, any myocardial infarction, any revascularization
Stent thrombosis by ARC definition | at 6 months, 9 months, 12 months, 24 months after procedure
Retenosis rate | at 9 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Principal Investigator — Department of Cardiology, First Affiliated Hospital of Air Force Medical University of Chinese PLA
Locations (1):
- Department of Cardiology, First Affiliated Hospital of Air Force Medical University of Chinese PLA, Xi'an, Shaanxi, China